CLINICAL TRIAL: NCT01519284
Title: A Double-blind, Randomised, Placebo- and Active-controlled Multiple-dose Study of BIA 9-1067 to Investigate Its Effect on Levodopa Pharmacokinetics Following a Levodopa/Carbidopa 100/25 mg Single-dose in Healthy Subjects
Brief Title: Study of BIA 9-1067 to Investigate Its Effect on Levodopa Pharmacokinetic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-114
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; entacapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Placebo Comparator): Placebo at all the dosing times
  Interventions: Drug: Placebo
- Group 2 (Experimental): Day 1 to 7:
  BIA 9-1067 5 mg: 7 AM dose Placebo: 8 AM; 4 PM; 12 PM dose
  Day 8:
  BIA 9-1067 5 mg: 7 AM dose Placebo+ levodopa/carbidopa 100/25 mg: 8 AM dose
  Interventions: Drug: BIA 9-1067 5 mg; Drug: Placebo; Drug: levodopa/carbidopa
- Group 3 (Experimental): Day 1 to 7:
  BIA 9-1067 15 mg: 7 AM dose Placebo: 8 AM; 4 PM; 12 PM dose
  Day 8:
  BIA 9-1067 15 mg: 7 AM dose Placebo+ levodopa/carbidopa 100/25 mg: 8 AM dose
  Interventions: Drug: Placebo; Drug: levodopa/carbidopa; Drug: BIA 9-1067 15 mg
- Group 4 (Experimental): Day 1 to 7:
  BIA 9-1067 30 mg: 7 AM dose Placebo: 8 AM; 4 PM; 12 PM dose
  Day 8:
  BIA 9-1067 30 mg: 7 AM dose Placebo + levodopa/carbidopa 100/25 mg: 8 AM dose
  Interventions: Drug: Placebo; Drug: levodopa/carbidopa; Drug: BIA 9-1067 30 mg
- Group 5 (Experimental): Day 1 to 7:
  Placebo: 7 AM dose; Entacapone 200 mg: 8 AM; 4 PM; 12 PM dose
  Day 8:
  Placebo: 7 AM dose Entacapone 200 mg + levodopa/carbidopa 100/25 mg: 8 AM dose
  Interventions: Drug: Entacapone; Drug: Placebo; Drug: levodopa/carbidopa

INTERVENTIONS:
Drug: BIA 9-1067 5 mg — BIA 9-1067 OPC, Opicapone 5 mg
  Other Names: OPC, Opicapone
  Arms: Group 2
Drug: Entacapone — Entacapone 200 mg
  Arms: Group 5
Drug: Placebo — placebo (four times a day)
  Other Names: PLC, placebo
Drug: levodopa/carbidopa — standard release levodopa/carbidopa 100/25 mg (single-dose)
  Arms: Group 2; Group 3; Group 4; Group 5
Drug: BIA 9-1067 15 mg — BIA 9-1067 OPC, Opicapone 15 mg
  Other Names: OPC, Opicapone
  Arms: Group 3
Drug: BIA 9-1067 30 mg — BIA 9-1067 OPC, Opicapone 30 mg
  Other Names: OPC, Opicapone
  Arms: Group 4

SUMMARY:
To investigate the effect of repeated dosing of BIA 9-1067 on the levodopa pharmacokinetics, in comparison to placebo and entacapone.

DETAILED DESCRIPTION:
Single-centre, double-blind, randomised, parallel-group study in 80 young male and female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Clinical laboratory test results clinically acceptable at screening and admission to the treatment period.
* Negative screen for alcohol and drugs of abuse at screening and admission to the treatment period.
* Non-smokers or ex-smokers for at least 3 months.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: intrauterine device (by the subject) and condoms (by the partner) or diaphragm (by the subject) and condoms (by the partner) or spermicide (by the subject) and condoms (by the partner).
* (If female) She had a negative urine pregnancy test at screening and admission to the treatment period.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* Any abnormality in the coagulation tests.
* Any abnormality in the liver function tests.
* A history of relevant atopy or drug hypersensitivity.
* A history or presence of narrow-angle glaucoma.
* A suspicious undiagnosed skin lesions or a history of melanoma.
* History of alcoholism or drug abuse.
* Consumed more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission to the treatment period.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to the treatment period.
* Had used non-selective monoamine oxidase (MAO) inhibitors within 2 weeks of admission to the treatment period.
* Had used medicines within 2 weeks of admission to the treatment period that may have affected the safety or other study assessments, in the investigator's opinion.
* Had previously received BIA 9-1067.
* Had used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Had participated in more than 2 clinical trials within the 12 months prior to screening.
* Had donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or had medical dietary restrictions.
* Cannot communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* Unwilling or unable to gave written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz-da-Silva, MD, PhD, Principal Investigator — BIAL - Portela & Cª S.A
Locations (1):
- Bial - Portela & Cª, S.A., S. Mamede Do Coronado, Portugal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started | 16 | 16 | 18 | 16 | 16
Completed | 16 | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Day 1 to 7:
  BIA 9-1067 5 mg: 7 AM dose Placebo: 8 AM; 4 PM; 12 PM dose
  Day 8:
  BIA 9-1067 5 mg: 7 AM dose Placebo+ levodopa/carbidopa 100/25 mg: 8 AM dose
  BIA 9-1067 5 mg: BIA 9-1067 OPC, Opicapone 5 mg
  Placebo: placebo (four times a day)
  levodopa/carbidopa: standard release levodopa/carbidopa 100/25 mg (single-dose)
- Group 3: Day 1 to 7:
  BIA 9-1067 15 mg: 7 AM dose Placebo: 8 AM; 4 PM; 12 PM dose
  Day 8:
  BIA 9-1067 15 mg: 7 AM dose Placebo+ levodopa/carbidopa 100/25 mg: 8 AM dose
  Placebo: placebo (four times a day)
  levodopa/carbidopa: standard release levodopa/carbidopa 100/25 mg (single-dose)
  BIA 9-1067 15 mg: BIA 9-1067 OPC, Opicapone 15 mg
- Group 4: Day 1 to 7:
  BIA 9-1067 30 mg: 7 AM dose Placebo: 8 AM; 4 PM; 12 PM dose
  Day 8:
  BIA 9-1067 30 mg: 7 AM dose Placebo + levodopa/carbidopa 100/25 mg: 8 AM dose
  Placebo: placebo (four times a day)
  levodopa/carbidopa: standard release levodopa/carbidopa 100/25 mg (single-dose)
  BIA 9-1067 30 mg: BIA 9-1067 OPC, Opicapone 30 mg
- Group 5: Day 1 to 7:
  Placebo: 7 AM dose; Entacapone 200 mg: 8 AM; 4 PM; 12 PM dose
  Day 8:
  Placebo: 7 AM dose Entacapone 200 mg + levodopa/carbidopa 100/25 mg: 8 AM dose
  Entacapone: Entacapone 200 mg
  Placebo: placebo (four times a day)
  levodopa/carbidopa: standard release levodopa/carbidopa 100/25 mg (single-dose)
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 16 | 16 | 18 | 16 | 16 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 18 | 16 | 16 | 82
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 9 | 8 | 8 | 41
  Male | 8 | 8 | 9 | 8 | 8 | 41

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration of Levodopa
Description: Cmax - Maximum plasma concentration of levodopa following a single oral administration of Sinemet® 100/25 on Day 8, and 5 mg, 15 mg and 30 mg BIA 9-1067 once-daily (QD), 200 mg entacapone thrice-daily (TID), and placebo, for 8 days
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng/mL | 1076 (292.7) | 1106 (420.3) | 943 (325.3) | 981 (488.5) | 928 (245)

2. Secondary Outcome: Tmax - Time to Reach Maximum Plasma Concentration of Levodopa
Description: Tmax - Time to Reach maximum plasma concentration of levodopa following a single oral administration of Sinemet® 100/25 on Day 8, and 5 mg, 15 mg and 30 mg BIA 9-1067 once-daily (QD), 200 mg entacapone thrice-daily (TID), and placebo, for 8 days.
Time Frame: 8 days
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
hours | 0.75 [0.25 to 1.0] | 0.75 [0.25 to 1.0] | 0.75 [0.25 to 3.0] | 0.75 [0.25 to 1.0] | 0.75 [0.25 to 1.0]

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve (AUC) of Levodopa From Time Zero to the Last Sampling Time at Which the Drug Concentration Was at or Above the Lower Limit of Quantification.
Description: AUC0-t - Area under the plasma concentration-time curve (AUC) of levodopa from time zero to the last sampling time following a single oral administration of Sinemet® 100/25 on Day 8, and 5 mg, 15 mg and 30 mg BIA 9-1067 once-daily (QD), 200 mg entacapone thrice-daily (TID), and placebo, for 8 days
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng.h/mL | 1578 (320.3) | 1785 (574.8) | 2102 (569.6) | 2202 (605.6) | 2146 (538.6)

4. Secondary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve (AUC) of Levodopa From Time Zero to Infinity
Description: AUC0-∞ - Area under the plasma concentration-time curve (AUC) of levodopa from time zero to infinity.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng.h/mL | 1649 (313.3) | 1873 (571.3) | 2233 (578.3) | 2381 (623.8) | 2253 (540.7)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 1/17 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/16 | 9/16 | 10/17 | 12/16 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=16) | Group 2 (N=16) | Group 3 (N=17) | Group 4 (N=16) | Group 5 (N=16)
spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=16) | Group 2 (N=16) | Group 3 (N=17) | Group 4 (N=16) | Group 5 (N=16)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Edema eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Application site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 0 | 0 | 0 | 1 | 0
Device breakage (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
CK increased (Investigations) | 0 | 1 | 0 | 2 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 2 | 2 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 3 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Menstrual discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes